CLINICAL TRIAL: NCT00372918
Title: An Interdisciplinary Interpretation of Transnasal Esophagoscopy Findings
Brief Title: Interpretation of Transnasal Esophagoscopy Findings
Acronym: TNE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Michael F. Vaezi, MD, PhD, MS epi, Vanderbilt University Medical Center Department of GI Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 060713
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Larynx Disease
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Transnasal Esophagoscopy
  Interventions: Procedure: Transnasal Esophagoscopy

INTERVENTIONS:
Procedure: Transnasal Esophagoscopy — fiberoptic exam of esophagus thru nares

SUMMARY:
The purpose of this study is to determine the prevalence of esophageal pathology in patients with voice disorders. In addition, , the intra- and interdisciplinary variability regarding the identification of esophageal pathology will be analyzed in this study.

DETAILED DESCRIPTION:
Throat symptoms are common complaints for many patients. Some symptoms are thought to be attributable to laryngopharyngeal reflux (i.e. the reflux of stomach acid to the level of the larynx). It is unclear what role laryngopharyngeal reflux (LPR) has in producing throat symptoms and its relationship to laryngeal pathology. LPR may be more carefully diagnosed if knowledge could be obtained regarding the presence of esophageal manifestations of reflux of stomach acid. Although LPR may occur in the absence of esophageal manifestations, the presence may make this diagnosis more probable. If so, therapy can be more carefully directed.

Using a flexible endoscope, otolaryngologists perform transnasal flexible laryngoscopy. This requires only topical anesthesia and occurs in the clinic setting. The small caliber transnasal esophagoscope was developed in recent years and is performed in a similar manner. It can provide key information regarding esophageal pathology. This obviates the need for administration of anesthesia (i.e. other than the topical, non-sedating agent). Transnasal flexible laryngoscopy is considered to be the standard of care for evaluation of the larynx. Transnasal esophagoscopy is an extension of this standard of care.

There are a number of studies demonstrating the safety and utility of transnasal esophagoscopy in humans. Typically these studies are composed of retrospectively on a select group of patients. Additionally the TNE findings are reviewed by one medical discipline. This study will be the first prospective analysis of TNE in which the findings will be reviewed in a multidisciplinary manner (i.e. otolaryngologists and gastroenterologist). Also, the population involved will be more general than previous studies, representing a myriad of throat symptoms.

ELIGIBILITY:
Inclusion criteria:

* Study participants include persons 18 years and older
* Patients presenting to the Vanderbilt Voice Center and complaining of throat symptoms. These include hoarseness, throat clearing/pain/burning, heartburn, globus sensation, and acidic/sour taste.
* New and return patients will be included.

Exclusion criteria:

* Participants who are unwilling to undergo the study
* Patients who have had prior esophagoscopy
* Those who do not sign the consent
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The intraobserver variability of Transnasal Esophagoscopy | one week apart
The interdisciplinary variability of Transnasal Esophagoscopy | one week apaart

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD PhD MS, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt ENT Clinic, Nashville, Tennessee, United States